CLINICAL TRIAL: NCT06779890
Title: Effect of Volatile-based Versus Total Intravenous Anesthesia on Cerebral Homeostasis and Neucognitive Function in Patients Undergoing Elective Craniotomy for Brain Tumor Excision.
Brief Title: Effect of Volatile- Based Versus Total Intravenous Anesthesia on Brain Homeostasis and Neurocognitive Outcome
Acronym: TIVolBrain
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Georgia Tsaousi (Other)
Responsible Party: Sponsor-Investigator, Georgia Tsaousi, Professor, Aristotle University Of Thessaloniki
Organization: Aristotle University Of Thessaloniki (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TIVAVolaBrain
Record Dates: First submitted 2025-01-08; First posted 2025-01-17 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Brain Edema Caused by Drugs; Cerebral Oxygenation
Keywords: sevoflurane; desflurane; total intravenous anesthesia; brain edema; brain oxygenation; neurocognitive outcome
MeSH Terms: conditions — Brain Edema | interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Total intravenous anesthesia in brain tumor surgery (Active Comparator): Propofol will be administered at concentrations maintaining BIS 40-60 up to surgery completion.
  Interventions: Drug: Sevoflurane; Drug: Desflurane
- Sevoflurane in brain tumor surgery (Experimental): Sevoflurane will be administered at concentrations maintaining MAC= 0.8 for the first 60 minutes , MAC=1.2 for the next 60 minutes and MAC= 0.8 until surgery completion.
  Interventions: Drug: Desflurane
- Desflurane in brain tumor surgery (Experimental): Desflurane will be administered at concentrations maintaining MAC= 0.8 for the first 60 minutes , MAC=1.2 for the next 60 minutes and MAC= 0.8 until surgery completion.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane will be administered at concentrations maintaining MAC= 0.8 for the first 60 minutes , MAC=1.2 for the next 60 minutes and MAC= 0.8 until surgery completion.
  Arms: Desflurane in brain tumor surgery; Total intravenous anesthesia in brain tumor surgery
Drug: Desflurane — Desflurane will be administered at concentrations maintaining MAC= 0.8 for the first 60 minutes , MAC=1.2 for the next 60 minutes and MAC= 0.8 until surgery completion.
  Other Names: Suprane
  Arms: Sevoflurane in brain tumor surgery; Total intravenous anesthesia in brain tumor surgery

SUMMARY:
The brain is a metabolic active organ with constant energy demands. Brain oxygen supply is secured via cerebral circulation. Brain tumor surgery is commonly associated with the tumor's underlying pathophysiology including brain swelling or edema. During craniotomy for brain tumor resection maintenance of cerebral hemodynamic stability is of paramount importance. Neuroinflammation is also a normal response to trauma, such as in the case of brain tumor surgery. The role of neuroinflammation in postoperative brain function is well documented and the aim is to limit it through an appropriate anesthetic approach.

Anesthetic agents used during surgery affect brain homeostasis. The anesthetic agent of choice for neurosurgery should deliver smooth and hemodynamically stable anesthesia, good operating conditions, and allow early neurological assessment. Also, the ideal anesthetic agent should preserve cerebral perfusion and neuroprotection.

The two most common categories of anesthetic agents used nowadays for elective craniotomy are intravenous and inhalational agents.

Propofol is the intravenous anesthetic agent of choice. The action of propofol involves a positive modulation of the inhibitory function of the neurotransmitter gamma-aminobutyric acid (GABA). Propofol causes a decrease in cerebral metabolic rate (CMR), intracranial pressure (ICP), cerebral perfusion pressure (CPP), and cerebral blood flow (CBF). It also is known for its antiemetic properties.

Volatile agents commonly used in neuroanesthesia clinical practice are sevoflurane and desflurane. Both of these agents decrease CMR while maintaining stable CPP. CBF alteration is dose-dependent. Desflurane evokes a greater cerebral vasodilation effect than sevoflurane. Sevoflurane is a well-known neuroprotective anesthetic agent traditionally used in neurosurgery. Both desflurane and sevoflurane are associated with early emergence.

Thus, this study aimed to explore the effect of volatile-based versus total intravenous anesthesia on cerebral homeostasis and neurocognitive function in patients undergoing elective craniotomy for brain tumor excision aiming to provide a basis for clinical rational drug use in patients undergoing craniotomy resection of supratentorial lesions.

DETAILED DESCRIPTION:
Each participant will receive standard monitoring (ECG, SpO2, SBP, BIS, urine output, temperature). More detailed hemodynamic monitoring will be obtained by the Edwards Lifesciences ClearSight system (CO, CI, SV, SVI, SVV, SVR, SVRI), while the analgesic efficacy of remifentanil will be assessed by Nociception index (NOL) monitoring.

TCI Remifentanil and propofol 2 mg/kg bolus dose will be the agents of choice for induction in anesthesia and cisatracurium will be used for neuromuscular blockade for intubation, while maintenance of anesthesia will be either volatile-based (sevoflurane or desflurane in low flow anesthesia approach) or propofol-based (TCI mode).

Protective mechanical ventilation will be chosen (7ml/kg IBW) with a respiratory rate to obtain a PaCO2 of 35-40 mmHg. PEEP will be changed for the best PaO2/FiO2 ratio and FiO2 of choice will be 0.5.

The radial artery catheterization will be applied for direct blood pressure measurement and arterial blood gas sampling (pH, PaO2, PaCO2, HCO3, BE, osmolality, lactic acid, Hb, glucose, Na and K will be measured).

The jugular bulb ipsilateral to the craniotomy site will be catheterized for receiving blood samples for blood gas analysis. The following oxygenation and metabolic parameters / derivates will be registered or calculated: SjvO2, pH, PjvO2, PjvCO2, HCO3, BE, Osmolality, Lactic acid jv, Hb, Glucose, Na, K, AjvDO2, AjvCO2, O2ERbr, eRQbr, AjvDL, and LOI.

Phases

* T0: after jugular bulb cannulation
* T30: 30 minutes after administration of either sevoflurane, desflurane, or propofol
* T60: 60 minutes after administration of either sevoflurane, desflurane, or propofol
* T120: 120 minutes after administration of either sevoflurane, desflurane, or propofol
* Τ180: 180 minutes after administration of either sevoflurane, desflurane, or propofol
* End of surgical procedure Phases TO, T30, T60, T180 and end of surgical procedures will be obtained with MAC= 0.8 for both volatile agents.

Phase T120 will be obtained with MAC= 1.2 for both volatile agents.

Blood samples for measuring S-100b, UCH-L1, GFAP will be obtained at phases T0, 6 hours, and 24 hours after administration of either sevoflurane, desflurane, or propofol Intraoperative consumption of volatile agents (sevoflurane or desflurane), propofol, and remifentanil will also be recorded.

Upon the opening of the dura matter the level of brain relaxation will be rated on a four-point scale (1. Completely relaxed, 2 sufficiently relaxed, 3 firm brain, 4 bulging brain) both by anesthesiologists and surgeons.

Awakening profile and emergence from anesthesia will be evaluated by the time needed for eye opening, response to verbal command, and extubation after discontinuation of administration of the anesthesia agent.

The Aldrete scoring system will be used for postanesthetic recovery assessment 30, 120 and 180 minutes during PACU stay. The Aldrete Scoring system consists of 5 clinically relevant parameters: muscle activity, respiration, circulation, consciousness and oxygen saturation.

Apfel score will be used for postoperative nausea and vomiting prediction. Any medication administered on PACU will be noted.

Recovery will be evaluated using two different scales. The Glasgow Outcome Scale- Extended (GOSE) assessment of global disability and recovery after traumatic brain injury will be applied both after PACU and hospital discharge. The quality of recovery- 40 is a 40-item questionnaire (QoR- 40) and will take place 24 hours postoperative and on discharge.

Neurocognitive testing will be performed at pre-anesthetic assessment, and 1 week after surgery completion using the Μontreal Cognitive Assessment (MoCA) scale.

ELIGIBILITY:
Inclusion Criteria:

* ASA-PS 1-3 (American Society of Anesthesiologists Physical Status classification)
* Elective or semi-elective craniotomy for brain tumor resection
* Signed informed consent

Exclusion Criteria:

* History of craniotomy at the same site
* Morbid obesity
* Delirious person before surgery
* Cognitive disturbances
* Preoperative heart rate (HR) <45 beats/min or second or third degree AV block
* Treatment with a-methyldopa, clonidine or other a2-adrenergic agonist
* Pregnancy
* Liver or renal failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in jugular venous oxygen saturation | Time Frame: At baseline (start of propofol or sevoflurane or desflurane), 30 minutes, 60 minutes, 120 minutes, 180 minutes and at the end of surgical procedure
  Alterations in jugular venous oxygen saturation (%), after administration of sevoflurane or desflurane or propofol as anesthetic agent

SECONDARY OUTCOMES:
Changes in brain relaxation score | Before dura opening
  Alterations in BRS after administration of sevoflurane or desflurane or propofol as anesthetic agent
Changes in Μontreal Cognitive Assessment (MoCA) | Preoperatively and one week following the end of surgical procedure
  Alterations in Μontreal Cognitive Assessment (MoCA) after administration of sevoflurane or desflurane or propofol as anesthetic agent.
Changes in GFAP | End of surgical procedure and 24 hours postoperatively
  Alterations in GFAP (ng/ml) levels after administration of sevoflurane or desflurane or propofol as anesthetic agent.
Changes in UCH-L1 | Baseline, end of surgical procedure and 24 hours postoperatively
  Alterations in UCH-L1 (ng/ml) after administration of sevoflurane or desflurane or propofol as anesthetic agent
Changes in S-100b protein | Baseline, end of surgical procedure and 24 hours postoperatively
  Alterations in S-100b (μg/L) after administration of sevoflurane or desflurane or propofol as anesthetic agent.

OTHER OUTCOMES:
Changes in arterio-jugular oxygen difference (AjvDO2) | At baseline (start of propofol or sevoflurane or desflurane), 30 minutes, 60 minutes, 120 minutes, 180 minutes and at the end of surgical procedure
  Alterations in arterio-jugular oxygen difference (AjvDO2 [ml/dl]), after after administration of sevoflurane or desflurane or propofol as anesthetic agent
Changes in arterio-jugular carbon dioxide difference (AjvCO2) | At baseline (start of propofol or sevoflurane or desflurane), 30 minutes, 60 minutes, 120 minutes, 180 minutes and at the end of surgical procedure
  Alterations in arterio-jugular carbon dioxide difference (AjvCO2 [mmHg]), after administration of sevoflurane or desflurane or propofol as anesthetic agent
Changes in brain oxygen extraction ratio (O2Erbr) | At baseline (start of propofol or sevoflurane or desflurane), 30 minutes, 60 minutes, 120 minutes, 180 minutes and at the end of surgical procedure
  Alterations in brain oxygen extraction ratio (O2Erbr [%]), after administration of sevoflurane or desflurane or propofol as anesthetic agent
Changes in Q-40 | Up to hospital discharge
  Alterations in Q-40 after administration of sevoflurane or desflurane or propofol as anesthetic agent

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Tsaousi, Professor, Principal Investigator — Aristotle University Of Thessaloniki
Locations (2):
- Greece (2):
  - AHEPA University Hospital, Thessaloniki
  - Aristotle University of Thessaloniki, Thessaloniki

IPD SHARING:
Plan to Share IPD: No